CLINICAL TRIAL: NCT02503605
Title: Prospective Randomized Clinical Trial to Test the Efficacy of a Biosimilar Recombinant Follicle Stimulating Hormone (FSH)vs. Urinary FSH in an Oocyte Donation Program
Brief Title: Biosimilar Versus Urinary Gonadotropins
Acronym: BEMDON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IVI Madrid (Other)
Collaborators: IVI Bilbao (Other)
Responsible Party: Principal Investigator, Antonio Requena, MD, PhD, IVI Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504-MAD-024-AR
Record Dates: First submitted 2015-07-16; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Infertility
Keywords: Biosimilar; ovarian stimulation; oocyte donor
MeSH Terms: conditions — Infertility | interventions — Urofollitropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biosimilar recombinant FSH (Active Comparator): Under current practice, 65 participants will be stimulated with 150 international units (IU)/day biosimilar recombinant FSH, .Daily doses of 0.25 miligrams gonadotropin-releasing hormone (GnRH) antagonist will start on day 6 of stimulation. From this day may also vary the dose of recombinant FSH biosimilar according ovarian response. In the presence of 3 or more follicles ≥17 mm, a single dose of 0.1 miligram GnRH agonist will be administered for triggering final oocyte maturation
  Interventions: Drug: Biosimilar recombinant FSH
- Urinary FSH (Active Comparator): Under current practice, 65 participants will be stimulated with 150 IU/day of urinary FSH. Daily doses of 0.25 miligrams gonadotropin-releasing hormone (GnRH) antagonist will start on day 6 of stimulation From this day may also vary the dose of urinary FSH according ovarian response. In the presence of 3 or more follicles ≥17 mm, a single dose of 0.1 miligram GnRH agonist will be administered for triggering final oocyte maturation
  Interventions: Drug: Urinary FSH

INTERVENTIONS:
Drug: Biosimilar recombinant FSH — Controlled ovarian stimulation with 150 IU/day biosimilar recombinant FSH
  Other Names: Bemfola
  Arms: Biosimilar recombinant FSH
Drug: Urinary FSH — Controlled ovarian stimulation with 150 IU/day urinary FSH
  Other Names: Fostipur
  Arms: Urinary FSH

SUMMARY:
Biosimilar drug marketing of recombinant FSH for the treatment of infertility is another step in simplifying fertility treatments, making them easier to manage and more accessible to patients. Taking in mind these arguments ,the study is proposed for determining equivalence in terms of biological effectiveness of an ovarian stimulation protocol with biosimilar recombinant FSH stimulation protocol vs. urinary FSH in oocyte donation program.

DETAILED DESCRIPTION:
Biosimilar products are drugs "like" biotechnological origin to other innovative biological medicines and that can be marketed once the patent has expired. These drugs are intended to achieve the same therapeutic benefit as biological medicinal resembles.

Because of the similarity in both the active substance in the formulation, it is intended to demonstrate the equivalence between the biosimilar medicine of recombinant FSH and FSH of urinary origin in terms of fitness.

The investigators' main objective is to perform a non-inferiority trial of biosimilar recombinant FSH product compared to a conventional ovarian stimulation protocol with urinary FSH in relation to the number of oocytes retrieved and the number of metaphase II oocytes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-35 years who meet the criteria for entry into the oocyte donor program and that are going to undergo controlled ovarian stimulation

Exclusion Criteria:

* Patient with a basal antral count> 20 follicles in total or <6 antral follicles per ovary
* Patients with comorbidities that, in the opinion of the investigator, may interfere with the treatment of ovarian stimulation
* The presence of ovarian cysts that judgment of the investigator would interfere with the stimulation or may pose a risk to the donor
* BMI <18 kg / m2
* BMI> 30 kg / m2
* Severe hypersensitivity to drugs with similar structure

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of metaphase II oocytes | 1 day

SECONDARY OUTCOMES:
Days of treatment | 2 weeks
Total dose of gonadotropins (IU) | 2 weeks
Estradiol concentration the day of human chorionic gonadotropin (hCG) administration (picograms/mililiterl) | 1 day
Progesterone concentration the day of hCG administration (nanograms/mililiter) | 1 day
Fertilization rate | 1 day
Percentage of cryopreserved embryos | 2 weeks
Implantation rate | 2 weeks
Cancellation rate | 1 week
Degree of satisfaction (numbers 0-10) | 1 month
Apoptosis rate in granulosa cells | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Requena, Md, PhD, Principal Investigator — IVI Madrid
Locations (1):
- IVI Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Background] Rettenbacher M, Andersen AN, Garcia-Velasco JA, Sator M, Barri P, Lindenberg S, van der Ven K, Khalaf Y, Bentin-Ley U, Obruca A, Tews G, Schenk M, Strowitzki T, Narvekar N, Sator K, Imthurn B. A multi-centre phase 3 study comparing efficacy and safety of Bemfola((R)) versus Gonal-f((R)) in women undergoing ovarian stimulation for IVF. Reprod Biomed Online. 2015 May;30(5):504-13. doi: 10.1016/j.rbmo.2015.01.005. Epub 2015 Jan 27. PMID 25735918
- [Background] Wolzt M, Gouya G, Sator M, Hemetsberger T, Irps C, Rettenbacher M, Vcelar B. Comparison of pharmacokinetic and safety profiles between Bemfola((R)) and Gonal-f((R)) after subcutaneous application. Eur J Drug Metab Pharmacokinet. 2016 Jun;41(3):259-65. doi: 10.1007/s13318-015-0257-6. Epub 2015 Jan 30. PMID 25633239